CLINICAL TRIAL: NCT01854541
Title: Visual Management for the Radiotherapy Process
Acronym: VMRTP
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: Maastro Clinic, The Netherlands (Other)
Responsible Party: Sponsor
Other Study IDs: VMRTP
Record Dates: First submitted 2013-05-13; First posted 2013-05-15 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Cancer
Keywords: Cancer; Radiotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radiotherapy: All patients receiving radiotherapy

SUMMARY:
The Visual Management for Radiotherapy Practice (VMRTP) aims to analyze, predict, visualize and shorten the waiting times for radiotherapy patients. The hypothesis is that this can be done by the introduction of models that can predict a patient being at risk for waiting too long as well as visual management tools that visualize the radiotherapy process.

DETAILED DESCRIPTION:
In a retrospective cohort of radiotherapy patients, time stamps of various steps in the radiotherapy process (diagnosis, multi-disciplinary board, referral, intake, simulation, treatment planning, quality control, first fraction of radiotherapy) will be collected. These will be combined with patient, tumor and patient-process (e.g. referring physician, treating physician, busy-at-the-time, referring hospital) related features. Based on these a predictive model will be learned that can estimate the probability at various stages of the process that the patient waits too long. Visual management will be developed that can visualize the predicted waiting time.

Process interventions aimed at reducing waiting times will be tested prospectively.

ELIGIBILITY:
Inclusion Criteria:

Patients receiving radiotherapy

Exclusion Criteria:

Patients not receiving radiotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated with radiotherapy
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2013-03; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
referral and first day of radiotherapy | 3 months
  Waiting time between referral and first day of radiotherapy

SECONDARY OUTCOMES:
Diagnosis and first day of radiotherapy | 3 months
  Waiting time between diagnosis and first day of radiotherapy
multi-disciplinary board and first day of radiotherapy | 3 months
  Waiting time between multi-disciplinary board and first day of radiotherapy
intake and first day of radiotherapy | 3 months
  Waiting time between intake and first day of radiotherapy
simulation and first day of radiotherapy | 3 months
  Waiting time between simulation and first day of radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- MAASTRO clinic, Maastricht, Netherlands